CLINICAL TRIAL: NCT05335070
Title: Non-randomized Prospective Pilot Study on Effect of Temporo-masseteric Nerve Block (TMNB) on Pain Reduction Following Wisdom Molar Extractions
Brief Title: Reducing Pain From Wisdom Molar Extractions
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Gayathri Subramanian, Associate Professor, Rutgers, The State University of New Jersey
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro2021002543
Record Dates: First submitted 2022-04-13; First posted 2022-04-19 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Acute Pain
Keywords: Temporo-masseteric Nerve Block; Twin Block; Prescription opioids; Acute Post-extraction pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Intervention Model Description: Prospective single-arm pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Temporo-masseteric Nerve Block (TMNB) Injection with Local Anesthetic (Experimental): Following lower third molar extraction under intravenous sedation, the patient will receive the TMNB local anesthetic nerve block using the standard dental local anesthetic, i.e,. 2% lidocaine with 1:100,000 epinephrine, on the side/s of lower wisdom molar extraction/s
  Interventions: Drug: Temporo-masseteric Nerve Block

INTERVENTIONS:
Drug: Temporo-masseteric Nerve Block — Following lower third molar extraction under intravenous sedation, the patient will receive the TMNB local anesthetic nerve block using the standard dental local anesthetic, i.e,. 2% lidocaine with 1:100,000 epinephrine on the side/s of the lower wisdom molar (third molar) extraction/s

SUMMARY:
This is a pilot study evaluating the ability of the Temporo-masseteric Nerve Block local anesthetic injection (this was called the Twin Block earlier) to reduce pain experienced by individuals undergoing removal of lower third molar(s) under intravenous sedation. Study participants will be queried for pain experience and pain medications taken during the first post-operative week and will present for a follow-up visit on Day 8.

DETAILED DESCRIPTION:
Each year, over 3.5 million, mostly, healthy young adults, have their third molar teeth ('wisdom teeth') removed under sedation and are often given opioid prescriptions for managing their pain. Wisdom molar removal is one of the most common reasons for opioid prescriptions to be given to adolescents. There is a national thrust to reduce both the dose and the duration of such opioid prescriptions because even short-term opioid exposures increase risk for narcotic addiction and misuse. Non-opioid options to manage pain will still allow for sufficient pain control without risking addiction, and hence, a fundamental component of our response to combat the current national opioid crisis.

The investigators are going to study a promising option- the Temporo-masseteric Nerve Block (TMNB) dental anesthetic injection (This was called the Twin Block earlier). The TMNB involves injecting the standard dental numbing medication in a way that 'numbs' the 'jaw-clencher' muscles on the side of the face. The investigators found that the TMNB relieved jaw pain stemming from these muscles, in a quick and sustained manner, even in patients whose pain following wisdom tooth removal primarily came from 'taut' and tender jaw-clencher muscles.

In this pilot study, the investigators will deliver the Temporo-masseteric Nerve Block (TMNB) injection to 20 individuals (study participants) who undergo extraction of at least 1 lower wisdom molar dental extraction under intravenous sedation, on the side/s of lower molar removal at the end of the procedure. The participant's pain experience, medications taken for pain, as well as any adverse effects from either pain medications or the TMNB injection will be queried for a period of 1 week following the procedure (remotely). On Day 8 (one week after the procedure), the participants will return for a follow-up visit. The participants' pain experience will be compared with historical controls. This study can support a simple, safe and inexpensive means to reduce pain after a common procedure and will provide proof-of-concept for the potential non-opioid analgesic role of TMNB injection following wisdom molar removal.

The participant will be advised to take a combination of ibuprofen and acetaminophen (600 mg ibuprofen and 325 mg acetaminophen) every 4-6 hours for pain, unless it is mild, for which OTC strength analgesics would prove adequate (ibuprofen or acetaminophen). 5/300 mg hydrocodone with acetaminophen will be utilized for pain management if the patient's pain does not respond to 600 mg ibuprofen and 325 mg acetaminophen, even an hour after medication.

The key outcomes collected will include peak-pain by 4 hours post-procedure (measured using numerical pain rating scale score NRS, from 0-10, with 0 corresponding to no pain, 1-3 corresponding to mild, 4-6 to moderate and 7-10 to severe pain), passive mouth opening, masticatory muscle pain to palpation (masseter and temporalis muscles), total dosage of pain medication/s consumed. Adverse effects to pain medication consumption (nausea/ drowsiness/ gastritis etc) or to the TMNB injection will also be recorded. Daily pain experience will be recorded each of the 7 days post-operatively either as a survey emailed to the participant or queried over the phone by research personnel.

A week after the procedure, the participant will present for a post-operative evaluation. The extraction/s site/s will be evaluated for any infection/delayed healing.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years of age or older (up to 64 years)
* Any demographic
* ASA 1 and 2 (mild or absent systemic illnesses, deemed fit for undergoing dental extractions under intravenous sedation)
* Not pregnant (as will not qualify to undergo procedure under intravenous sedation as part of routine standard-of-care)
* Adequate mental ability to understand and provide informed consent
* Has smart phone and internet connection

Exclusion Criteria:

* Age older than 64 years (because they are poor candidates for undergoing procedures under intravenous sedation)
* Pregnant
* Incapable of providing informed consent
* Any systemic condition that renders the patient at higher risk for complications under intravenous sedation
* Documented allergy to the dental local anesthetic
* Inability to tolerate any of the commonly used pain medications such as combination opioids, acetaminophen (Tylenol®) or ibuprofen (Motrin® or Advil®)
* Limitation in adequate mouth opening in presence/absence of pain

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-09-13 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Peak post-operative Pain Score | up to 4 hours on day of procedure, post-procedure
  Every 30 minutes, the patient's pain score (Numerical Pain Rating Scale with scores from 0-10, (the NRS scale), with 0= no pain, 1-3= mild pain, 4-6= moderate pain, 7-10= severe pain) will be recorded to document peak pain score by hour 4. If the patient were to report a score from 7-10 at any time, no additional delay/pain score enquiry will take place and the patient will be directed to take the first dose of post-operative pain medication as described elsewhere.
Mean Numerical Pain Rating Scale pain score | One week
  The average pain score reported by the patient during the entire post-operative week will be assessed
Passive Mouth opening | Baseline, post-procedure (Day 1) and at post-operative visit (Day 8)
  Passive mouth opening will be measured (in mm) at baseline, post-procedure before as well as 15 min after TMNB injection and finally, during the post-operative visit (Day 8) will be measured
Masticatory muscle pain to palpation- Temporalis and Masseter | Baseline, post-procedure (Day 1) and at post-operative visit (Day 8)
  Numerical pain rating scale pain scores reported by the patient upon palpation of the masseter and temporalis muscles will be recorded at baseline, post-procedure (before and 15 min after TMNB injection) and at the post-operative visit one week after procedure
Total dose of pain medication- acetaminophen, ibuprofen and hydrocodone | 8 Days
  Total dose of pain medications consumed over the first post-operative week, for each of the medications will be recorded in mg
Adverse effects | 8 days
  The patient will be queried each day for any adverse effects from pain medications and any adverse effects at the site of injection (infection, pain etc)

CONTACTS AND LOCATIONS:
Overall Officials: Gayathri D Subramanian, PhD, DMD, Principal Investigator — Rutgers School of Dental Medicine
Locations (1):
- The University Hospital- Dental Clinic, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
After anonymizing, IPD will be shared after the study is completed.
Supporting Information: Study Protocol
Time Frame: After study completion, upon review of request
Access Criteria: A written request will be evaluated and responded to.

REFERENCES:
- [Background] Quek SYP, Gomes-Zagury J, Subramanian G. Twin Block in Myogenous Orofacial Pain: Applied Anatomy, Technique Update, and Safety. Anesth Prog. 2020 Jun 1;67(2):103-106. doi: 10.2344/anpr-67-01-03. PMID 32633773
- [Background] Kanti V, Ananthan S, Subramanian G, Quek SYP. Efficacy of the twin block, a peripheral nerve block for the management of chronic masticatory myofascial pain: A case series. Quintessence Int. 2017 Oct 6:725-729. doi: 10.3290/j.qi.a39094. Online ahead of print. PMID 28990015
- [Background] Quek S, Young A, Subramanian G. The twin block: a simple technique to block both the masseteric and the anterior deep temporal nerves with one anesthetic injection. Oral Surg Oral Med Oral Pathol Oral Radiol. 2014 Sep;118(3):e65-7. doi: 10.1016/j.oooo.2014.01.227. Epub 2014 Feb 6. PMID 24703404